CLINICAL TRIAL: NCT07010874
Title: THE EFFECT OF REMOTE NURSING INTERVENTIONS BASED ON THE EMPOWERMENT PROCESS MODEL ON PEOPLE WITH DEMENTIA AND THEIR FAMILY CAREGIVERS: A MIXED METHODS STUDY
Brief Title: THE EFFECT OF REMOTE NURSING INTERVENTIONS BASED ON THE EMPOWERMENT PROCESS MODEL ON PEOPLE WITH DEMENTIA AND THEIR FAMILY CAREGIVERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Naile Bilgili, Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GaziU-Aysun ERDAL
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Dementia of Alzheimer Type
Keywords: dementia caregiver; remote nursing; caregiving burden; web-based

STUDY DESIGN:
Intervention Model Description: This study was designed as a mixed methods research. In the quantitative part of this study, it was planned as a randomized controlled pretest-posttest (parallel) study to evaluate the effect of remote nursing interventions based on the empowerment model on individuals with dementia and family caregivers. After the completion of the quantitative part of the qualitative part of the study, in-depth semi-structured interviews will be conducted to determine the experiences and opinions of individuals with dementia and family caregivers regarding remote nursing interventions based on the empowerment model.
Who Masked: Outcomes Assessor
Masking Description: The list of participants for the study will be obtained from the Alzheimer's Social Life Center. The nurse working at the center will create a list of eligible individuals by evaluating caregivers and dementia patients according to the criteria for participation in the study. The list will be forwarded to the independent researcher and the participants will be randomly assigned to the intervention and control groups using the simple random randomization method with the list produced by the independent researcher from the https://www.randomizer.org/ web page.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The intervention for this group will last 10 weeks and will be conducted in weekly sessions. The empowerment process model was adopted to guide the intervention process. Distance nursing interventions based on the model will be carried out through a web page called "Take Care of Yourself". Each participant will have a unique username and password so that their login details and frequency of visits to the website will be recorded. During the 10-week intervention period, caregivers will be provided with 8 modules of training content.
  Interventions: Other: REMOTE NURSING INTERVENTIONS BASED ON THE EMPOWERMENT PROCESS MODEL
- control (No Intervention): Dementia patients and their relatives in the control group will continue to receive standard services provided by the Alzheimer's Social Life Center.

INTERVENTIONS:
Other: REMOTE NURSING INTERVENTIONS BASED ON THE EMPOWERMENT PROCESS MODEL — The duration of the intervention is determined as 10 weeks. Distance nursing interventions based on the model will be carried out through a web page called "Take Care of Yourself". Each participant will have a unique username and password while using the website, so that login information and the frequency of visiting the website will be recorded. During the 10-week intervention period, caregivers will be provided with 8 modules of training content. In the first session of the intervention, the website will be introduced, personal goals will be set and the session will be completed with the planning of the next week. personal goals will be set, and in the last session of the intervention, feedback will be given to the individuals by the researcher regarding the achievement of their personal goals and their ability to cope with future difficulties.
  Arms: intervention

SUMMARY:
In this study, it is planned to evaluate the effect of remote nursing interventions based on the empowerment model on individuals with dementia and family caregivers. It was designed as a mixed method research. It chose explanatory sequential mixed methods design as a mixed method type. The research will be conducted at the Alzheimer's Social Life Center affiliated to Ankara Metropolitan Municipality between June 01 and December 31, 2025. The quantitative part of the study was planned in a randomized controlled pretest-posttest (parallel) study design. The study will be conducted with 30 caregivers in the intervention group and 30 in the control group. Descriptive Information Form, Zarit Care Burden Scale, Caregiver Readiness Scale, Mini Mental Test and NPE - Neuropsychiatric Inventory will be used as data collection tools. The intervention period was determined as 10 weeks. Remote nursing interventions based on the model will be carried out through the web page named "Take Care of Yourself". Dementia patients and their relatives in the control group will continue to receive standard services provided by the Alzheimer Social Life Center. One week after the end of the intervention, the data collection tools will be applied again by the nurse at the center to the dementia patients and caregivers in both groups. Quantitative data will be evaluated using appropriate statistics in SPSS 23.0 package program. After the quantitative part of the study is completed, the qualitative part will be applied. The qualitative part was designed in a descriptive phenomenological design. In-depth individual interviews will be conducted with individuals who meet the inclusion criteria. A semi-structured interview form will be used in individual interviews. When it is decided that data saturation has been reached, the data collection phase of the research will be terminated. Data analysis will be carried out with the content analysis approach. The data will be analyzed using the MAXQDA 20 program. After the data collected from the qualitative and quantitative phases are analyzed separately, the findings of the two phases will be integrated in the interpretation phase.

DETAILED DESCRIPTION:
In the study, the intervention will be carried out in weekly sessions. A empowerment process model has been adopted to guide the intervention process. Prior to the study, a pilot study will be conducted at a different Alzheimer's Social Life Centre with dementia caregivers who meet the study participation criteria in order to test the usability of the developed website and determine the comprehensibility of the content of the training modules prepared for the maintenance process.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older,
* Are literate,
* Are able to use the internet,
* Have a close relative diagnosed with dementia related to Alzheimer's disease and are in the early stages of dementia (Mini Mental Test score between 19 and 24).
* Informal caregivers who have been providing care to a person with dementia for at least 6 months will be included in the study.

Exclusion Criteria:

* Individuals with physical (vision and hearing impairments) or psychological (schizophrenia, bipolar disorder, intellectual disabilities, etc.) conditions that prevent them from using the program,
* Caregivers of individuals with dementia diagnosed with Alzheimer's disease, who also have a life-threatening illness (central nervous system infections, organic brain damage, COPD, cancer, etc.) that increases the care burden and are currently undergoing active treatment for this illness,
* Caregivers of individuals with dementia who live in long-term care facilities or multiple homes and do not have a primary caregiver will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Zarit Car Burden Scale | It will be applied before the start of the program and 15 days after its completion.
  Scale, developed by Zarit and Zarit in 1990, has a Cronbach's alpha value of 0.91. The validity and reliability of the Turkish version were established by Özer, Yurttaş, and Akyıl (2012). It consists of 18 statements that determine the impact of caregiving on an individual's life. The scale is evaluated based on the total score. The score range is 0-72. A higher score indicates a higher caregiving burden.
Preparedness for Caregiving Scale | It will be administered before the start of the program and 15 days after its completion.
  Scale was developed by Archbold and Stewart (1986). Its validity and reliability for the Turkish society were established by Karaman and Karadakovan (2015). . The scale consists of eight items and an additional item that asks caregivers about the area in which they would like to be better prepared to provide care.

SECONDARY OUTCOMES:
NPE - Neuropsychiatric Inventory | It will be administered before the start of the application and 15 days after the end of the application.
  Turkish standardization and validity reliability study was conducted in 2005. It is conducted retrospectively (up to the last month) in the form of an interview with a person who is in daily contact with the patient and has witnessed the patient's behavior. Symptoms of NPE include: delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, abnormal motor behaviors, sleep/nighttime behaviors, and changes in appetite/eating.
Mini Mental Test | It will be administered before the start of the application and 15 days after the end of the application.
  This test will be used to assess the cognitive health of dementia patients.It will also be used to identify participants who are in the early stages of dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Metropolitan Municipality Alzheimer's Social Life Center, Ankara, YENİMAHALLE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] World Health Organization (2023). Dementia. Erişim Tarihi: 02 Aralık 2023, Erişim Adresi: https://www.who.int/news-room/fact-sheets/detail/dementia.
- [Result] Yeh J, Pond B, Beld M, Garcia A, Mauricio J, Mata-Pacheco J, Eldridge C, Ross L. Enhancing Dementia Knowledge and Self-Efficacy of In-Home Supportive Services Caregivers Through Online Training. J Appl Gerontol. 2023 Apr;42(4):617-626. doi: 10.1177/07334648221144023. Epub 2022 Dec 9. PMID 36482678
- [Result] Widyastuti, R. H., Sahar, J., Rekawati, E., & Kekalih, A. (2024). Development of Online Training Modules on Dementia Care at Home for Family Caregivers. The Open Nursing Journal, 18(1).
- [Result] Salehinejad, S., Jannati, N., Azami, M., Mirzaee, M., & Bahaadinbeigy, K. (2024). A web-based information intervention for family caregivers of patients with Dementia: a randomized controlled trial. Journal of Information Science, 50(1), 104-115.
- [Result] Pinyopornpanish M, Pinyopornpanish K, Soontornpun A, Tanprawate S, Nadsasarn A, Wongpakaran N, Wongpakaran T. Perceived stress and depressive symptoms not neuropsychiatric symptoms predict caregiver burden in Alzheimer's disease: a cross-sectional study. BMC Geriatr. 2021 Mar 12;21(1):180. doi: 10.1186/s12877-021-02136-7. PMID 33711938
- [Result] Hong QX, Wang WF, Yang YH, Tung YC, Dai HJ, Hsu WC, Huang LC, Jhang KM. The effectiveness of virtual passport, an app-based intervention, for dementia care. Front Psychiatry. 2024 Sep 26;15:1457923. doi: 10.3389/fpsyt.2024.1457923. eCollection 2024. PMID 39391088
- [Result] Gómez-Morales, A., Coon, D. W., Glinka, A., Stirling, R., Pipe, T., Joseph, R. P., Garcia-Segura, S. (2023). Training alternatives for Alzheimer's disease and related dementia caregivers: Assessing economic and environmental benefits of internet of health things. Journal of Cleaner Production, 418, 138206.
- [Result] Coon DW, Gomez-Morales A. Modifiable Risk Factors for Brain Health and Dementia and Opportunities for Intervention: A Brief Review. Clin Gerontol. 2023 Mar-Apr;46(2):143-154. doi: 10.1080/07317115.2022.2114396. Epub 2022 Aug 22. PMID 35996225
- [Result] Christie HL, Dam AEH, van Boxtel M, Kohler S, Verhey F, de Vugt ME. Lessons Learned From an Effectiveness Evaluation of Inlife, a Web-Based Social Support Intervention for Caregivers of People With Dementia: Randomized Controlled Trial. JMIR Aging. 2022 Dec 7;5(4):e38656. doi: 10.2196/38656. PMID 36476485
- [Result] Biliunaite I, Kazlauskas E, Sanderman R, Truskauskaite-Kuneviciene I, Dumarkaite A, Andersson G. Internet-Based Cognitive Behavioral Therapy for Informal Caregivers: Randomized Controlled Pilot Trial. J Med Internet Res. 2021 Apr 7;23(4):e21466. doi: 10.2196/21466. PMID 33825687
- [Result] Bauernschmidt D, Hirt J, Langer G, Meyer G, Unverzagt S, Wilde F, Wittmann J, Bieber A. Technology-Based Counselling for People with Dementia and Their Informal Carers: A Systematic Review and Meta-Analysis. J Alzheimers Dis. 2023;93(3):891-906. doi: 10.3233/JAD-221194. PMID 37125549
- [Result] Bastoni S, Wrede C, da Silva MC, Sanderman R, Gaggioli A, Braakman-Jansen A, van Gemert-Pijnen L. Factors Influencing Implementation of eHealth Technologies to Support Informal Dementia Care: Umbrella Review. JMIR Aging. 2021 Oct 8;4(4):e30841. doi: 10.2196/30841. PMID 34623314
- [Result] Andrews JS, Desai U, Kirson NY, Enloe CJ, Ristovska L, King S, Birnbaum HG, Fleisher AS, Ye W, Kahle-Wrobleski K. Functional limitations and health care resource utilization for individuals with cognitive impairment without dementia: Findings from a United States population-based survey. Alzheimers Dement (Amst). 2016 Dec 9;6:65-74. doi: 10.1016/j.dadm.2016.11.005. eCollection 2017. PMID 28229124
- [Result] Alzheimer's Association. (2023). 2023 Alzheımer's Dısease Facts and Fıgures Erişim Tarihi: 02 Kasım 2023, Erişim Adresi: https://www.alz.org/media/Documents/alzheimers-facts-and-figures.pdf
- [Result] Akça-Kalem, S., Hanağası, H., Cummings, J. L., & Gürvit, H. (2005, September). Validation study of the Turkish translation of the Neuropsychiatric Inventory (NPI). In 21st international conference of Alzheimer's Disease İnternational, Sept (p. 47).
- [Result] Adriani, D., Imran, Y., Mawi, M., Amani, P., & Ilyas, E. I. (2020). Effect of Brain Gym® exercises on cognitive function and brain-derived neurotrophic factor plasma level in elderly: a randomized controlled trial. Universa Medicina, 39(1), 34-41.